CLINICAL TRIAL: NCT03616132
Title: A Prospective, Non-randomized, Open-label, Non-comparative, First-in-Man Study to Evaluate the Feasibility and Safety of Sirolimus-eluting Iron Bioresorbable Coronary Scaffold System
Brief Title: A First-in-Man Study to Evaluate the Feasibility and Safety of Sirolimus-eluting Iron Bioresorbable Coronary Scaffold System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBS-FIM-MY
Record Dates: First submitted 2018-07-30; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-07

CONDITIONS: Single Coronary Vessel Disease

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBS implantation (Experimental): Implantation of IBS in patients with coronary artery lesions.
  Interventions: Device: Device: Sirolimus-eluting Iron Bioresorbable Coronary Scaffold System

INTERVENTIONS:
Device: Device: Sirolimus-eluting Iron Bioresorbable Coronary Scaffold System — Implantation of Sirolimus-eluting Iron Bioresorbable Coronary Scaffold System (IBS)

SUMMARY:
The study is a pilot clinical trial for Sirolimus-eluting Iron Bioresorbable Coronary Scaffold System（IBS）. The main purpose of this study is to evaluate the feasibility, preliminary safety and efficacy of IBS. To provide the basis for subsequent large-scale, multi-center, randomized controlled clinical trials of IBS.

DETAILED DESCRIPTION:
* A prospective, non-randomized trial
* Study population: 15 patients
* Clinical follow up will be required at postoperative, 1 month, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years;
* All the subjects perform the angiography, Intra-vascular ultrasound (IVUS) and Optical coherence tomography (OCT) at 1 year and 3 years.
* The primary study endpoint is target lesion failure (TLF) at 1 month post procedure; and imaging findings as the secondary study endpoint. To evaluate the feasibility, safety and performance of IBS.

ELIGIBILITY:
Inclusion Criteria:

* All patients participating in this clinical trial must meet the following criteria:

  1. Age of 18-75， males or non pregnancy females;
  2. Subject must have evidence of myocardial ischemia (e.g., stable, unstable angina, post-infarct angina or silent ischemia) suitable for elective PCI;
  3. One target lesion, and target lesion can be completely covered by a single stent;
  4. Target lesion length ≤ 18 mm, target lesion diameter between 3.0 mm to 3.5 mm (visual);
  5. Visual assessment of target lesion stenosis ≥70%, TIMI blood flow≥ 1;
  6. Subject who understand the purpose of testing, voluntary and informed consent, patients undergoing invasive imaging follow-up.

Exclusion Criteria:

* Patients will be excluded if any of the following conditions apply:

General:

1. Within 1 week of any acute myocardial infarction or myocardial enzymes did not return to normal;
2. Implantation of stent in target vessel within 1 year , patients with planned intervention again within six months;
3. Patients who performed coronary artery bypass (coronary artery bypass grafting);
4. Patients with contraindications for coronary artery bypass graft surgery;
5. Severe heart failure (NYHA class III and above) or left ventricular ejection fraction<40% (ultrasonic or left ventricular angiography);
6. Preoperative renal function: serum creatinine > 2.0 mg/dl or 177 mu mol/L; receiving hemodialysis;
7. Patients have ischemic stroke half a year before implantation, patients have transient ischemic attack 3 months before implantation, patients have high coagulation tendency judged by investigator or laboratory examination;
8. Bleeding, active gastrointestinal ulcers, brain hemorrhage or subarachnoid hemorrhage, contraindications on antiplatelet agents and anticoagulant therapy; patients would not allow to undergoing antithrombotic therapy;
9. Aspirin, clopidogrel, heparin, contrast agent, poly lactic acid polymer, rapamycin and metal allergies;
10. Patients who have a history of disease related to iron overload or iron disorder, such as hereditary hemochromatosis, etc;
11. The patient's life expectancy is less than 12 months;
12. Patient participated in other drug or medical device study and does not meet the primary study endpoint in clinical trials time frame;
13. Poor compliance and patients unable to complete the study in accordance with the requirements;
14. Patient with heart transplant;
15. The unstable arrhythmia, such as high risk ventricular extra systole and ventricular tachycardia;
16. Cancer needs chemotherapy;
17. Patients of immune suppression, autoimmune diseases, planned or undergoing immunosuppressive therapy;
18. Planning or being receiving long-term anticoagulant therapy, such as heparin, warfarin, etc;
19. With six months for elective surgery requires stop using aspirin and clopidogrel;
20. Blood test prompted platelet count < 100 x 109/L, or > 700 x 109/L, white blood cells < 3 x 109/L, or abnormal liver function (ALT、AST 3 times greater than normal range);
21. Patients with diffuse peripheral vascular disease; cannot use 6F catheter;
22. Patients with valvular surgery in the past.

Exclusion criteria by angiography:

1. Chronic total occlusion (TIMI blood flow=0 before implantation) , left main coronary artery lesion, ostial lesion, multiple vessel lesion, branch lesion and bridge lesion which branch vessel diameter ≥ 2.0 mm (if the ostium of branch vessel stenosis >40% or needs balloon predilation); visible thrombus in target vessels;
2. Severe calcified lesions and distorted disease which unable to predilation, lesion not suitable for stent delivery and expansion;
3. In-stent restenosis;
4. Myocardial bridge is involved in target lesion;
5. In order to reach the target lesion, study stent has to go through the previous implanted stent;
6. Predilation balloon can't expand completely in target lesion site, judgment standard for fully expansion as below, patients are excluded when do not meet any item:

A. DS% < 40%（visual），highly recommend DS% ≤20% B. TIMI blood flow= class 3（visual） C. No angiography complications (e.g., distal embolization, lateral branch closed) D. No interlining level NHLBI type D - F E. No continuous chest pain (> 5 minutes), and F. No lower or higher ST segment >5 minutes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-03-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Study Device related Composite Endpoint (Target Lesion Failure) | 1 month after implantation
  Target Lesion Failure is defined as the composited endpoints of including cardiac death, Target vessel related myocardial infarction (TV-MI) and clinical indicated target lesion revascularization (CI-TLR), also known as MACE (major adverse cardiac events).

SECONDARY OUTCOMES:
Immediate Success Rate | Immediate postoperative
  1. Device Success:
     Successfully transit and release the IBS at target lesion, then withdraw the delivery system. Immediate residual stenosis < 30% and TIMI blood flow is class 3 (visual).
  2. Lesion Success: Any method of intervention therapy, the residual stenosis of the target lesion < 30% and TIMI blood flow is class 3(visual).
Clinical Success | Hospitalized period postoperative within 7 days
  Defined as based on lesion success, there is no major adverse cardiac events in the hospitalization period.
Performance Evaluation of IBS | Immediate postoperative
  4 class (Excellent, good, general, bad) to evaluate the push ability, performance of through the lesions, performance of cover the lesions, support force, withdraw ability.
Device related Composite Endpoint (DoCE) | 6 Month, 1 Year, 2 Years, 3 Years, 4 Years, 5 Years postprocedure
  Target Lesion Failure, defined as the composited endpoints of including cardiac death, Target vessel related myocardial infarction (TV-MI) and clinical indicated target lesion revascularization (CI-TLR), also known as MACE (major adverse cardiac events).
Patient related Clinical Composite Endpoint (PoCE) | 30 Days, 6 Months, 1 Year, 2 Years, 3 Years, 4 Years, 5 Years postprocedure
  Including all-cause mortality, all myocardial infarction and target lesion revascularization.
Stent Thrombosis defined by ARC | Acute(0-24 hours), Subacute(24 hours-30 days), Late(30 days-1 year),Very late(after 1 year)
  Timing (acute, sub-acute, late and very late) Evidence (definite and probable)
Acute stent retraction | Immediate postoperative
  Angiographic Endpoint
In-stent, in-segment, proximal and distal minimum lumen diameter (MLD) | Immediate postoperative, 1 year, 3 years
  Angiographic Endpoint
In-stent, in-segment, proximal and distal Diameter stenosis(DS) | 1 year, 3 years
  Angiographic Endpoint
In-stent, in-segment, proximal and distal Late lumen loss (LLL) | 1 year, 3 years
  Angiographic Endpoint
In-stent, in-segment, proximal and distal Angiographic defined restenosis (ABR) | 1 year, 3 years
  Angiographic Endpoint
Vasomotion | 1 year, 3 years
  Defined as the average diameter change of lumen diameter before and after using nitroglycerin.
Analysis of Morphometric, lesion composition and scaffold strut data obtained with OCT | : Immediate postoperative, 1 year, 3 years
  Optical Coherence Tomography Endpoint
Analysis of Vascular and scaffold morphology obtained with IVUS | Immediate postoperative,1 year, 3 years
  Intra-Vascular Ultrasound Endpoint

CONTACTS AND LOCATIONS:
Locations (2):
- Malaysia (2):
  - Institut Jantung Negara, Kuala Lumpur, Negeri Selangor
  - University Malaya Medical Centre, Kuala Lumpur, Negeri Selangor